CLINICAL TRIAL: NCT00724854
Title: Evaluation of Rapid Virological Response in HCV Patients Treated With PegIntron and Ribavirin - APEGIN Trial
Brief Title: Evaluation of Rapid Virologic Response Among HCV Patients Treated With PegIntron and Rebetol in Brazil (Study P05427)
Acronym: APEGIN
Status: Completed | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: P05427; 001/05
Record Dates: First submitted 2008-07-25; First posted 2008-07-30 (Estimated); Results first posted 2011-01-10 (Estimated); Last update posted 2015-02-25 (Estimated); Status verified 2015-02

CONDITIONS: Hepatitis C, Chronic; Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C | interventions — peginterferon alfa-2b; Ribavirin

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Mono-infected with HCV: Participants infected with Hepatitis C Virus (HCV).
  Interventions: Biological: PegIntron (peginterferon alfa-2b; SCH 54031); Drug: Rebetol (ribavirin; SCH 18908)
- Co-infected with HCV and HIV: Participants co-infected with HCV and Human Immunodeficiency Virus (HIV).
  Interventions: Biological: PegIntron (peginterferon alfa-2b; SCH 54031); Drug: Rebetol (ribavirin; SCH 18908)

INTERVENTIONS:
Biological: PegIntron (peginterferon alfa-2b; SCH 54031) — PegIntron administered in accordance with approved labeling
  Other Names: SCH 54031
Drug: Rebetol (ribavirin; SCH 18908) — Rebetol administered in accordance with approved labeling
  Other Names: SCH 18908

SUMMARY:
The objective of the study is to evaluate, in each group, the number of participants who achieve rapid virological response (RVR) after 4 weeks treatment with PegIntron and Rebetol. The study will also assess whether RVR is a reliable predictor of sustained virologic response (defined as undetectable viral load at 24 weeks post-treatment).

ELIGIBILITY:
Inclusion Criteria:

* Willing to participate in the study and sign the Informed Consent Form
* Established HCV infection, confirmed by molecular biology test (positive qualitative polymerase chain reaction [PCR] test)
* Can be treatment-naïve, have retreatment, or co-infected with HIV
* Be under treatment with PegIntron in combination with ribavirin, starting up to 14 days before the screening visit

Exclusion Criteria:

* Participants who have not confirmed their willingness to participate in the study or have refused to sign the Free and Informed Consent Form
* Prior treatment with PegIntron (combined with ribavirin or not)
* History of alcohol abuse in the past 6 months
* Decompensated liver disease
* Severe heart disease
* Decompensated thyroid disorder
* Neoplasia
* Type 1 diabetes mellitus - uncontrolled or hardly controlled
* Seizures - uncontrolled
* Primary immune deficiency
* Men and women not using appropriate contraceptive methods
* Pregnancy or lactation
* For participants co-infected with HIV: HIV-related opportunistic disease in the past 6 months or CD4 count lower than 200 cells/mm^3

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants infected with Hepatitis C Virus (HCV) who are undergoing treatment with PegIntron and Rebetol in accordance with approved labeling at approximately 60 sites in Brazil. Participants could be treatment-naïve, undergoing re-treatment, or co-infected with Human Immunodeficiency Virus (HIV).
Sampling Method: Probability Sample
Enrollment: 1146 (Actual)
Dates: Start 2006-08; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

REFERENCES:
- [Result] Santos C, Reis A, Dos Santos CV, Damas C, Silva MH, Viana MV, Ferraz ML, Carnauba D, El-Far F, Serra F, Diaz RS. The use of real-time PCR to detect hepatitis C virus RNA in dried blood spots from Brazilian patients infected chronically. J Virol Methods. 2012 Jan;179(1):17-20. doi: 10.1016/j.jviromet.2011.06.012. Epub 2011 Jun 24. PMID 21871496

RESULTS

PARTICIPANT FLOW:
Groups:
- Mono-infected With HCV: Participants infected with Hepatitis C Virus (HCV), received PegIntron plus Rebetol, administered in accordance with approved labeling.
- Co-infected With HCV and HIV: Participants co-infected with Hepatitis C Virus (HCV) and Human Immunodeficiency Virus (HIV), received PegIntron plus Rebetol, administered in accordance with approved labeling.
Period: Overall Study
Arm/Group | Mono-infected With HCV | Co-infected With HCV and HIV
Started | 1010 (Number enrolled was 1146. 64 participants were screen failures.) | 72 (Number enrolled was 1146. 64 participants were screen failures.)
Completed | 607 | 41
Not Completed | 403 | 31
Not completed — Lack of Efficacy | 187 | 13
Not completed — Lost to Follow-up | 87 | 10
Not completed — Adverse Event | 62 | 4
Not completed — Other | 42 | 3
Not completed — Death | 11 | 0
Not completed — Change of treatment | 7 | 0
Not completed — Withdrawal by Subject | 5 | 0
Not completed — Adverse event + lack of efficacy | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mono-infected With HCV | Co-infected With HCV and HIV | Total
Number analyzed (Participants) | 1010 | 72 | 1082
Age, Customized [Number; unit: Participants]
  <=40 years | 193 | 36 | 229
  >40 years | 817 | 36 | 853
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 444 | 23 | 467
  Male | 566 | 49 | 615
Region of Enrollment [Number; unit: participants]
  Brazil | 1010 | 72 | 1082

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Rapid Virologic Response After 4 Weeks of Treatment
Description: Rapid virologic response (RVR) was defined as Hepatitis C Virus Ribonucleic acid (HCV RNA) negative after 4 weeks of treatment.
Time Frame: Assessed at Treatment Week 4
Measure: Number; unit: Participants
Arm/Group | Mono-infected With HCV | Co-infected With HCV and HIV
Number analyzed (Participants) | 1010 | 72
Participants | 551 | 32

2. Secondary Outcome: Number of Participants Who Achieved Sustained Virologic Response (SVR)
Description: SVR was defined as non-detectable HCV RNA 24 weeks post-treatment.
Time Frame: Assessed at 24 weeks post-treatment
Measure: Number; unit: Participants
Arm/Group | Mono-infected With HCV | Co-infected With HCV and HIV
Number analyzed (Participants) | 1010 | 72
Participants | 375 | 24

3. Secondary Outcome: Number of Participants With RVR Who Also Achieved SVR
Description: RVR was defined as HCV RNA negative after 4 weeks of treatment. SVR was defined as non-detectable HCV RNA 24 weeks or more post-treatment.
Time Frame: Assessed at Treatment Week 4 (RVR) and 24 weeks post-treatment (SVR)
Population: Participants who achieved RVR at Treatment Week 4.
Measure: Number; unit: Participants
Arm/Group | Mono-infected With HCV | Co-infected With HCV and HIV
Number analyzed (Participants) | 551 | 32
Participants | 300 | 19

4. Secondary Outcome: Assessment of Response at Treatment Week 48 for Genotypes 2 and 3, and Treatment Week 72 for Genotypes 1, 4, and 5, in Participants With RVR
Description: Participants who achieved RVR at Treatment Week 4 who were considered to have SVR (non-detectable HCV RNA at Treatment Week 48 for genotypes 2 and 3, and Treatment Week 72 for genotypes 1, 4, and 5). Participants from the Mono-infected with HCV group and the Co-infected with HCV and HIV group, were identified as either Genotype 1, 2, 3, 4, or 5.
Time Frame: Treatment Week 48 and Treatment Week 72
Population: Participants who achieved RVR at Treatment Week 4.
Measure: Number; unit: Participants
Arm/Group | Mono-infected With HCV | Co-infected With HCV and HIV
Number analyzed (Participants) | 551 | 32
Participants
  No SVR | 251 | 13
  SVR | 300 | 19

5. Secondary Outcome: Assessment of Baseline Characteristics in Participants With SVR
Description: Baseline characteristics assessed were age, gender, and genotype.
Time Frame: 24 Weeks post-treatment
Population: Participants with SVR
Measure: Number; unit: Participants
Arm/Group | Mono-infected With HCV | Co-infected With HCV and HIV
Number analyzed (Participants) | 375 | 24
Participants
  Age <=40 years | 75 | 11
  Age >40 years | 300 | 13
  male | 203 | 17
  female | 172 | 7
  Genotype 1 | 247 | 14
  Genotype non-1 | 128 | 10

ADVERSE EVENTS:
Arm/Group | Mono-Infected With HCV | Co-Infected With HCV and HIV | Not Evaluated
Serious Adverse Events (participants affected / at risk) | 52/1010 | 0/72 | 8/64
Other Adverse Events (participants affected / at risk) | 762/1010 | 61/72 | 42/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mono-Infected With HCV (N=1010) | Co-Infected With HCV and HIV (N=72) | Not Evaluated (N=64)
ANAEMIA (Blood and lymphatic system disorders) | 8 (8) | 0 (0) | 0 (0)
HAEMOLYTIC ANAEMIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
LEUKOPENIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
PANCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
ANGINA PECTORIS (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
CARDIAC FAILURE (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
HYPOACUSIS (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
RETINAL DETACHMENT (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 3 (3) | 0 (0) | 1 (1)
ASCITES (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1)
DIARRHOEA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2)
FAECALOMA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
HAEMATEMESIS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
MELAENA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
OESOPHAGEAL ULCER HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
OESOPHAGEAL VARICES HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
PERITONITIS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
STOMATITIS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
UPPER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
VOMITING (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
ASTHENIA (General disorders) | 1 (1) | 0 (0) | 0 (0)
DEATH (General disorders) | 2 (2) | 0 (0) | 0 (0)
FATIGUE (General disorders) | 1 (1) | 0 (0) | 0 (0)
MALAISE (General disorders) | 1 (1) | 0 (0) | 0 (0)
MULTI-ORGAN FAILURE (General disorders) | 1 (1) | 0 (0) | 0 (0)
PYREXIA (General disorders) | 1 (1) | 0 (0) | 1 (1)
CHOLELITHIASIS (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
CHOLESTASIS (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
JAUNDICE (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0)
APPENDICITIS (Infections and infestations) | 4 (4) | 0 (0) | 0 (0)
CELLULITIS (Infections and infestations) | 1 (4) | 0 (0) | 0 (0)
CENTRAL NERVOUS SYSTEM ABSCESS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
PNEUMONIA (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
PULMONARY TUBERCULOSIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
SEPSIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
UROSEPSIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
INJURY (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
DIABETES MELLITUS (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
DIABETIC KETOACIDOSIS (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
METABOLIC ACIDOSIS (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
COLON CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
ASTERIXIS (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
DIZZINESS (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
ENCEPHALOPATHY (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
HEPATIC ENCEPHALOPATHY (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0)
OPTIC NEURITIS (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
QUADRIPLEGIA (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
CONFUSIONAL STATE (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
DEPRESSION (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2)
RENAL FAILURE (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
RENAL FAILURE ACUTE (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
INTERSTITIAL LUNG DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0) | 0 (0)
PRURITUS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
LEG AMPUTATION (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
DEEP VEIN THROMBOSIS (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
HYPOTENSION (Vascular disorders) | 2 (2) | 0 (0) | 0 (0)
THROMBOPHLEBITIS (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mono-Infected With HCV (N=1010) | Co-Infected With HCV and HIV (N=72) | Not Evaluated (N=64)
ANAEMIA (Blood and lymphatic system disorders) | 165 (171) | 18 (19) | 5 (6)
LEUKOPENIA (Blood and lymphatic system disorders) | 38 (39) | 6 (6) | 1 (1)
NEUTROPENIA (Blood and lymphatic system disorders) | 59 (60) | 7 (9) | 5 (5)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 34 (34) | 5 (5) | 1 (1)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 63 (65) | 6 (6) | 3 (3)
DIARRHOEA (Gastrointestinal disorders) | 76 (77) | 8 (8) | 7 (8)
NAUSEA (Gastrointestinal disorders) | 122 (138) | 8 (11) | 6 (6)
VOMITING (Gastrointestinal disorders) | 42 (44) | 5 (5) | 2 (3)
ASTHENIA (General disorders) | 284 (309) | 14 (15) | 17 (17)
FATIGUE (General disorders) | 105 (110) | 9 (9) | 4 (4)
INFLUENZA LIKE ILLNESS (General disorders) | 132 (136) | 2 (2) | 9 (9)
IRRITABILITY (General disorders) | 99 (99) | 9 (9) | 2 (2)
MALAISE (General disorders) | 57 (58) | 5 (6) | 3 (3)
PYREXIA (General disorders) | 274 (292) | 33 (37) | 14 (15)
WEIGHT DECREASED (Investigations) | 72 (72) | 8 (8) | 1 (1)
ANOREXIA (Metabolism and nutrition disorders) | 126 (129) | 15 (15) | 7 (7)
DECREASED APPETITE (Metabolism and nutrition disorders) | 63 (68) | 7 (7) | 3 (3)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 78 (86) | 11 (12) | 0 (0)
MYALGIA (Musculoskeletal and connective tissue disorders) | 280 (302) | 33 (34) | 12 (12)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 32 (34) | 4 (4) | 4 (4)
DIZZINESS (Nervous system disorders) | 69 (71) | 3 (3) | 2 (2)
HEADACHE (Nervous system disorders) | 257 (295) | 19 (21) | 10 (10)
DEPRESSION (Psychiatric disorders) | 100 (100) | 9 (10) | 9 (9)
INSOMNIA (Psychiatric disorders) | 94 (95) | 4 (4) | 3 (3)
COUGH (Respiratory, thoracic and mediastinal disorders) | 84 (86) | 6 (6) | 3 (3)
ALOPECIA (Skin and subcutaneous tissue disorders) | 93 (93) | 8 (8) | 3 (3)
PRURITUS (Skin and subcutaneous tissue disorders) | 140 (146) | 6 (6) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Whenever a Principal Investigator wishes to use the results of the study, he/she should contact the sponsor to obtain the authorization.